CLINICAL TRIAL: NCT05129488
Title: 2 Hour Dispensing Evaluation of Biotrue ONEday Contact Lenses With EPG03 Packaging Solution Compared to Commercially Available Biotrue ONEday Contact Lenses
Brief Title: Biotrue ONEday Contact Lenses With EPG03 Packaging Solution Compared to Biotrue ONEday Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-005
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2022-11

CONDITIONS: Contact Lens Wearer

STUDY DESIGN:
Intervention Model Description: Approximately 30 habitual soft contact lens wearing subjects will be enrolled in this two-hour randomized, contralateral, double-masked (subject and investigator masked), repeated measures dispensing study.
Masking Description: The participant and investigator were masked and randomized allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All participants received Biotrue ONEday lenses with and without an alternate packaging solution (Experimental): Participants were given both Commercially available Biotrue ONEday lenses and Biotrue ONEday Contact Lenses with EPG03 Packaging Solution. Lens material is made from a hydrophilic copolymer of 2- hydroxyethyl methacrylate and N-vinylpyrrolidone and is 78% water by weight when immersed in saline solution. EPG03 Packaging Solution contains a phosphate buffered saline solution containing potassium chloride, poloxamine, poloxamer 181, glycerol (glycerin), erythritol, and polyquaternium-1.
  Interventions: Device: All participants received Biotrue ONEday lenses with and without an alternate packaging solution (EPG03)

INTERVENTIONS:
Device: All participants received Biotrue ONEday lenses with and without an alternate packaging solution (EPG03) — Participants were given both Commercially available Biotrue ONEday lenses and Biotrue ONEday Contact Lenses with EPG03 Packaging Solution. Lens material is made from a hydrophilic copolymer of 2- hydroxyethyl methacrylate and N-vinylpyrrolidone and is 78% water by weight when immersed in saline solution.EPG03 Packaging Solution contains a phosphate buffered saline solution containing potassium chloride, poloxamine, poloxamer 181, glycerol (glycerin), erythritol, and polyquaternium-1.

SUMMARY:
The objective of this 2 hour study is to evaluate the clinical performance of Biotrue ONEday lenses with an alternate packaging solution (EPG03) compared to commercially available Biotrue ONEday lenses. This novel contact lens packaging solution contains known elements in the ophthalmic industry and is safe for use.

DETAILED DESCRIPTION:
Approximately 30 habitual soft contact lens wearing subjects will be enrolled in this two-hour randomized, contralateral, double-masked (subject and investigator masked), repeated measures dispensing study. All subjects will be seen for a Screening/Dispensing Visit at which informed consent will be obtained and eligibility will be assessed. If subjects satisfy all eligibility criteria and none of the exclusion criteria, subjects will be dispensed study lenses according to unique randomization schedules that will be provided to each Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and have capacity to read, understand and provide written voluntary informed consent.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis.
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent.

Exclusion Criteria:

1. Participating in a conflicting study in the opinion of the Investigator.
2. Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Schafer, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch and Lomb Site 01, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- All Participants Received Biotrue ONEday Lenses With and Without an Alternate Packaging Solution: Participants were given both Commercially available Biotrue ONEday lenses and Biotrue ONEday Contact Lenses with EPG03 Packaging Solution. Lens material is made from a hydrophilic copolymer of 2- hydroxyethyl methacrylate and N-vinylpyrrolidone and is 78% water by weight when immersed in saline solution.EPG03 Packaging Solution contains a phosphate buffered saline solution containing potassium chloride, poloxamine, poloxamer 181, glycerol (glycerin), erythritol, and polyquaternium-1.
Period: Overall Study
Arm/Group | All Participants Received Biotrue ONEday Lenses With and Without an Alternate Packaging Solution
Started | 33; 66 Eyes (33 eyes (contralateral assignment))
Contact Lenses With Solution | 30; 60 Eyes
Contact Lenses Without Solution | 30; 60 Eyes
Completed | 30; 60 Eyes (All 3 subjects that did not complete reported at baseline corneal staining above the protocol limits. Neither test nor control articles were dispensed.)
Not Completed | 3; 6 Eyes
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Participants Received Biotrue ONEday Lenses With and Without an Alternate Packaging Solution (EPG03): Participants were given both Commercially available Biotrue ONEday lenses and Biotrue ONEday Contact Lenses with EPG03 Packaging Solution. Lens material is made from a hydrophilic copolymer of 2- hydroxyethyl methacrylate and N-vinylpyrrolidone and is 78% water by weight when immersed in saline solution.EPG03 Packaging Solution contains a phosphate buffered saline solution containing potassium chloride, poloxamine, poloxamer 181, glycerol (glycerin), erythritol, and polyquaternium-1.
Arm/Group | Participants Received Biotrue ONEday Lenses With and Without an Alternate Packaging Solution (EPG03)
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Normalized logMAR Visual Acuity
Description: logMAR visual acuity typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision. 0.02 is considered 1 letter on the chart Normalized logMAR VA is a change from baseline measurement. It is calculated by taking the logMAR VA from the baseline refraction (No contact lens) and subtracting the logMAR VA with the contact lens.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Biotrue ONEday Lenses With an Alternate Packaging Solution (EPG03): Biotrue ONEday Contact Lenses With EPG03 Packaging Solution lens material is made from a hydrophilic copolymer of 2- hydroxyethyl methacrylate and N-vinylpyrrolidone and is 78% water by weight when immersed in saline solution. EPG03 Packaging Solution contains a phosphate buffered saline solution containing potassium chloride, poloxamine, poloxamer 181, glycerol (glycerin), erythritol, and polyquaternium-1.
- Biotrue ONEday Lenses: Biotrue ONEday lenses: Commercially available Biotrue ONEday lenses
Arm/Group | Biotrue ONEday Lenses With an Alternate Packaging Solution (EPG03) | Biotrue ONEday Lenses
Number analyzed (Participants) | 30 | 30
LogMAR | -0.01 (0.070) | -0.02 (0.109)

ADVERSE EVENTS:
Time Frame: 2 hours
Groups:
- Biotrue ONEday Contact Lenses With EPG03 Packaging Solution: Biotrue ONEday Contact Lenses With EPG03 Packaging Solution lens material is made from a hydrophilic copolymer of 2- hydroxyethyl methacrylate and N-vinylpyrrolidone and is 78% water by weight when immersed in saline solution. EPG03 Packaging Solution contains a phosphate buffered saline solution containing potassium chloride, poloxamine, poloxamer 181, glycerol (glycerin), erythritol, and polyquaternium-1.
- Biotrue ONEday Contact Lenses: Commercially Available Biotrue ONEday Contact Lenses
Arm/Group | Biotrue ONEday Contact Lenses With EPG03 Packaging Solution | Biotrue ONEday Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT05129488/Prot_SAP_000.pdf